CLINICAL TRIAL: NCT00509626
Title: A Physical Activity Intervention to Prevent Weight Gain in Breast Cancer Patients
Brief Title: Physical Activity or Usual Care in Preventing Weight Gain in Women With Stage I or Stage II Breast Cancer Undergoing Chemotherapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: CDR0000555830; P30CA006927 (NIH); FCCC-FCRB-05-009
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Last update posted 2010-02-12 (Estimated); Status verified 2010-02

CONDITIONS: Breast Cancer; Depression; Fatigue; Psychosocial Effects of Cancer and Its Treatment; Weight Changes
Keywords: fatigue; psychosocial effects of cancer and its treatment; weight changes; depression; stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms; Depression; Fatigue; Body Weight Changes | interventions — Exercise Therapy; Psychiatric Rehabilitation

INTERVENTIONS:
Behavioral: exercise intervention
Other: questionnaire administration
Procedure: CAM exercise therapy
Procedure: management of therapy complications
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Physical activity may prevent or reduce weight gain in women receiving chemotherapy for early stage breast cancer.

PURPOSE: This randomized phase I/II trial is studying physical activity to see how well it works compared with usual care to prevent or reduce weight gain in women with stage I or stage II breast cancer undergoing chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility for conducting a clinical trial that uses a 6-month physical activity intervention initiated within 45 days after surgery for early-stage breast cancer and prior to initiation of adjuvant chemotherapy, hormonal therapy, and/or radiotherapy. (phase I)
* Determine if participation in a 6-month physical activity intervention initiated within 45 days after surgery for early-stage breast cancer decreases weight gain in patients treated with adjuvant chemotherapy. (phase II)
* Determine if participation in a 6-month physical activity intervention initiated within 45 days after surgery for early-stage breast cancer differentially affects weight change in women who are premenopausal compared to those who are postmenopausal at diagnosis. (phase II)

Secondary

* Determine if participation in a 6-month physical activity intervention initiated within 45 days after surgery for early-stage breast cancer decreases gains in adiposity in patients treated with adjuvant chemotherapy. (phase II)
* Determine if participation in a 6-month physical activity intervention initiated within 45 days after surgery for early-stage breast cancer differentially affects change in adiposity among women who are premenopausal compared to those who are postmenopausal at diagnosis. (phase II)
* Determine if participation in a 6-month physical activity intervention initiated within 45 days after surgery for early-stage breast cancer decreases the frequency of depressive symptomology and improves quality of life among patients treated with adjuvant chemotherapy. (phase II)

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating site and menopausal status (premenopausal vs postmenopausal). Patients are randomized to 1 of 2 intervention arms.

* Arm I (exercise and usual care): Patients receive usual care and are enrolled in an exercise and weight control program at Curves® fitness center. The Curves® program, which begins during the third week of study, uses aerobic activity and resistance training to reduce weight and increase strength and fitness. Patients exercise a minimum of 3 times per week, approximately 30 minutes every time, for up to 6 months in the absence of disease progression or unacceptable toxicity. Patients' physical activity is measured at baseline and at the 3- and 6-month follow-up visits.

Patients also undergo behavior modification counseling with a study nurse to help them overcome the specific barriers to adhering to the recommended exercise routine. Counseling sessions are conducted every 2 to 3 weeks during chemotherapy and at least monthly after completion of chemotherapy for up to 6 months, starting within 2 weeks after randomization and prior to initiation of the Curves® intervention.

* Arm II (control: usual care alone): Patients receive usual care and general advice on coping with their breast cancer treatment for up to 6 months in the absence of disease progression or unacceptable toxicity. Patients receive no counseling or recommendations concerning emotional and practical barriers encountered during breast cancer treatment.

Dietary information is obtained from patients by telephone during three 24-hour dietary recalls performed within 2 weeks of baseline and at the 3-month and 6-month follow-up visits to estimate total energy intake throughout the study. Patients complete questionnaires at baseline and periodically during study assessing demographic characteristics and established breast cancer risk factors, medical history, and health changes. Weight, adiposity as measured by waist circumference, quality of life, and depressive symptomology are assessed at baseline and at the 3- and 6-month follow-up visits.

After completion of the study intervention, patients are followed for up to 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Diagnosis of primary breast cancer

  * Newly diagnosed stage I or II disease
* Receiving care at a participating Fox Chase Cancer Center CCOP Research Base (FCRB) member site

  * Geisinger Clinic and Medical Center (phase I)
  * Main Line Health (phase I)
  * Any of the other participating FCRB member sites (phase II)
* Study intervention is scheduled to begin anytime after surgery up to 3 months after completion of adjuvant chemotherapy
* Treatment plan includes adjuvant chemotherapy
* Hormone receptor status not specified

Exclusion criteria:

* Treatment plan includes trastuzumab (Herceptin®) or bevacizumab
* Recurrent breast cancer

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Female
* Premenopausal or postmenopausal
* Has obtained medical clearance by oncologist and breast surgeon to participate in this study
* Body mass index ≥ 20 kg/m^2 and < 39 kg/m^2

Exclusion criteria:

* Hemoglobin < 12 g/dL
* ANC < 1,500/mm^3
* Any medical condition that restricts participation in a physical activity program (e.g., exercise-induced angina, uncontrolled hypertension, dementia, or a major psychological problem)
* Answers "yes" to any questions on the Physical Activity Readiness Questionnaire (PAR-Q) and PAR-Q not reviewed by a physician who subsequently approves participation in the physical activity intervention
* Known to be pregnant or breastfeeding
* Unwilling to commit or unable to participate in a 6-month physical activity intervention (unable to exercise, usually travels away from home overnight more than once per week, and/or has plans to be away from home for more than two weeks in the next 6 months)
* Previously diagnosed with another primary cancer other than basal cell or squamous cell carcinoma of the skin
* Exercising regularly prior to intervention (i.e., reports current participation in vigorous or moderate activity at least 3 days per week for at least 30 minutes each day on the International Physical Activity Questionnaire)
* Unable to speak and read English

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No neoadjuvant chemotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Accrual (phase I)
Retention (phase I)
Weight change after 6 months (phase II)

SECONDARY OUTCOMES:
Adiposity as measured by waist circumference at 3 and 6 months
Health-related quality of life as measured by the Short-Form Health Survey-12 Physical and Mental Component Summary scales
Depressive symptomology as measured by the Center for Epidemiologic Studies Depression Scale

CONTACTS AND LOCATIONS:
Overall Officials: Penny Anderson, MD, Study Chair — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania, United States